CLINICAL TRIAL: NCT06888232
Title: Safety and Efficacy of Immunomodulator Drug Thalidomide in Multi-transfused Thalassemia Patients: A Single Center Experience From South Punjab, Pakistan
Brief Title: Safety and Efficacy of Immunomodulator Drug Thalidomide in Multi-transfused Thalassemia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DRASLAMCHMULTAN
Record Dates: First submitted 2025-03-15; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Thalassemia
MeSH Terms: conditions — Thalassemia | interventions — Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thalidomide group (Experimental): Thalidomide was administered at a dose of 1.5 mg/kg/day, and all patients continued standard iron chelation therapy and other supportive treatments as per institutional protocols.
  Interventions: Drug: Thalidomide

INTERVENTIONS:
Drug: Thalidomide — Thalidomide was administered at a dose of 1.5 mg/kg/day, and all patients continued standard iron chelation therapy and other supportive treatments as per institutional protocols.

SUMMARY:
This study aimed to determine the safety and efficacy of thalidomide in multi-transfused thalassemic children.

DETAILED DESCRIPTION:
Given the significant burden of transfusion dependency, an effective and safe inducer is needed that could improve quality of life and reduce the healthcare costs associated with frequent transfusions and iron chelation therapy. If this study could establish the safety of thalidomide in terms of teratogenicity along with its efficacy, it would be a great support to multi-transfused thalassemic children.

ELIGIBILITY:
Inclusion Criteria:

* Children of both genders
* Aged 2-5 years
* With transfusion-dependent thalassemia (TDT)
* Whose parents/guardians showed willingness to adhere to follow-up visits

Exclusion Criteria:

* Children with uncontrolled infections
* Significant hepatic or renal dysfunction
* Malignancy
* Known contraindications to thalidomide

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of treatment | 6 months
  Efficacy was categorized as excellent response showing an increase in hemoglobin by 1-2 g/dL or freedom from blood transfusions, partial response as an increase in hemoglobin <1 g/dL or a decrease in transfusion frequency, or no response if there was no increase in hemoglobin or an increase in transfusion requirement within three months.
Safety of treatment | 6 months
  Treatment was considered safe if no adverse events were documented based on clinical assessment and laboratory findings.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Aslam, FCPS, Principal Investigator — Children's Hospital and institute of Child Health Multan, Punjab, Pakistan; Sara Rubab, FCPS, Principal Investigator — Children's Hospital and institute of Child Health Multan, Punjab, Pakistan
Locations (1):
- The Children's Hospital & Institute of Child Health, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared on a reasonable request.